CLINICAL TRIAL: NCT03477981
Title: Acceptability of Dietary Fibre-based Foods to Reduce Dietary Fat Uptake
Brief Title: Acceptability of Dietary Fibre-based Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Proposal v4 04JAN2010
Record Dates: First submitted 2017-10-27; First posted 2018-03-27 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants will consume their habitual diet with standard white bread for two week, then will be given the alginate bread for two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Other): Participants will receive standard white bread for two weeks and then alginate bread for two weeks. All participants will receive the bread in the same order.
  Interventions: Other: Alginate bread

INTERVENTIONS:
Other: Alginate bread — White bread with 4% alginate (wet weight of dough) included into the bread.

SUMMARY:
Obesity is a wide reaching problem in the United Kingdom. The most widely used obesity therapies are based around drugs that reduce dietary fat digestion, and thereby reduce uptake of calories from the diet. While such therapies have proved effective, patient compliance is low due to the unwanted gastrointestinal side effects of these drugs. Dietary fibre is generally classified as dietary material of plant origin that is indigestible to humans. Dietary fibre is in fact a wide range of different compounds that have varied effects on the human body. Initial findings from this laboratory suggest that some types of fibre can greatly reduce the rate that fat is digested and absorbed in the gut.

Whether such fibre-based test foods are acceptable (i.e. taste good, are easy to include in the diet and do not cause any unwanted gastrointestinal side effects) will be assessed in longer term studies. To carry these studies out, healthy adults will be recruited. Participants will attend an induction visit and will be asked to keep a food diary, and fill out daily questionnaires on general well-being and feelings of fullness over a two-week period whilst consuming the standard white bread given to them. Following this two-week period, participants will attend the study centre again. At this time, participants will be provided with dietary fibre-based study food (bread) to substitute into their standard diet over the following two weeks (further bread will be provided as and when required). Participants will fill out the same diaries and questionnaires as before over the first two week period.

DETAILED DESCRIPTION:
This study aims to test the acceptability of fibre-based foods in terms of their palatability, ease of incorporation into the diet and the lack of unwanted side effects of consumption. To meet these aims, participants will be provided with bread to incorporate into their diet (by substituting like-for-like) over a two-week period. During this time, participants will record what they have eaten, along with their general feelings of well-being throughout this period. These measures will be compared to the same data collected over the two-week period prior to giving the participants the study foods (as a "background" measure of food intake and general well-being).

To carry these studies out, healthy adults will be recruited. Participants will attend an induction visit at Newcastle University where we will take informed consent. Participants will then be asked to keep a food diary, and fill out daily questionnaires on their general well-being and feelings of fullness for the entirety of the following two weeks whilst consuming the standard white bread given to them. Following this two-week period, participants will attend the study centre again and will be provided with dietary fibre-based study food (breads) to substitute into their standard diet over the following two weeks (further foods will be provided as and when required). They will fill out the same diaries and questionnaires as they did before over the first two week period.

The wellbeing questionnaire will be filled out by participants every day with a more detailed questionnaire completed at the end of each week. Volunteers will complete the more detailed questionnaire five times. Once at the start of the study (baseline) and then at then once at the end of each week consuming standard white bread and once at the end of each week consuming the alginate bread. The standard wellbeing questionnaire will be completed every day the volunteers are on the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* over the age of 18

Exclusion Criteria:

* Individuals with a known allergy to any of the study foods
* Individuals who wish not to consume the study foods)
* Individuals who will not be able to consume their standard diet over the study period (e.g. due to holidays etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2012-01-18 (Actual); Study Completion 2012-01-18 (Actual)

PRIMARY OUTCOMES:
A change in side effects with consumption of alginate bread | Every day volunteers take part in the study (28 days)
  A change in the number gastrointestinal side effects described by the volunteers
A change in visual analogue scale (VAS) score of question: How have you been feeling today, alert or sleepy? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, fine or nauseous? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, full or starving? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, not bloated or bloated? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, not flatulent or flatulent? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, calm or irritable? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: How have you been feeling today, relaxed or anxious? | Measured once per day for 28 days
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.

SECONDARY OUTCOMES:
A change in visual analogue scale (VAS) score of question: Have you been suffering from; light-headedness or dizziness, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; Blurred Vision, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; a difficulty to concentrate, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; excessive thirst, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; headaches/migraines, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; cravings for sweets, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Have you been suffering from; abdominal discomfort, not at all or very? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Overall, how would you say the following have been: bowel habit, constipated or diarrhoea? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Overall, how would you say the following have been: urgency to pass stool, less than normal more than normal? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Overall, how would you say the following have been: abdominal pain or discomfort, no pain or terrible? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.
A change in visual analogue scale (VAS) score of question: Overall, how would you say the following have been: amount of flatulence, less than normal or more than normal? | Once per week at the end of each study week (4 weeks)
  Visual analogue scale (VAS) score between 0 - 10. The VAS scale is 10 cm long horizontal line and measured from the left hand side. The distance from the left hand side that the volunteer marks on the scale generates the score. The question relating to the scale will have a polar answer at each end of the VAS, as described in the title with the first answer on the left hand end and the second answer on the right hand end.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available